CLINICAL TRIAL: NCT03344172
Title: Randomized Phase II Trial of Pre-Operative Gemcitabine, Nab-Paclitaxel, and Hydroxychloroquine With or Without Avelumab (PGHA vs. PGH)
Brief Title: Pre-Operative Trial (PGHA vs. PGH) for Resectable Pancreatic Cancer
Acronym: 17-134
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Suspected Serious Adverse Events related to treatment
Sponsor: Nathan Bahary, MD (Other)
Collaborators: Pfizer (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Nathan Bahary, MD, associate professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC# 17-134; R01CA181450 (NIH)
Record Dates: First submitted 2017-10-03; First posted 2017-11-17 (Actual); Results first posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-04

CONDITIONS: Pancreatic Cancer Resectable
MeSH Terms: interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Hydroxychloroquine; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PGHA (Experimental): Gemcitabine, Nab-Paclitaxel, and hydroxychloroquine and Avelumab
  Interventions: Drug: Gemcitabine, Nab-Paclitaxel, hydroxychloroquine and Avelumab
- PGH (Experimental): Gemcitabine, Nab-Paclitaxel, and hydroxychloroquine
  Interventions: Drug: Gemcitabine, Nab-Paclitaxel, and hydroxychloroquine

INTERVENTIONS:
Drug: Gemcitabine, Nab-Paclitaxel, hydroxychloroquine and Avelumab — Days 1, 8, 15 of Cycles 1 and 2: gemcitabine (1000mg/m^2) and nab-paclitaxel (125mg/m^2) Beginning on Day 8 of Cycle 1: hydroxychloroquine (600mg/BID) daily until day of surgery Day 1 of Cycle 3: avelumab (10mg/kg)
  Other Names: PGHA
  Arms: PGHA
Drug: Gemcitabine, Nab-Paclitaxel, and hydroxychloroquine — Days 1, 8, 15 of Cycles 1 and 2: gemcitabine (1000mg/m^2) and nab-paclitaxel (125mg/m^2) Beginning on Day 8 of Cycle 1: hydroxychloroquine (600mg/BID) daily until day of surgery
  Other Names: PGH
  Arms: PGH

SUMMARY:
This is a randomized phase II trial that will examine the ability of Avelumab to improve the clinical activity of a pre-operative regimen of gemcitabine, nab-paclitaxel and hydroxychloroquine in subjects with potentially resectable adenocarcinoma of the pancreas.

DETAILED DESCRIPTION:
This is a phase II, non-blinded, adaptively randomized trial. Patients with PDA are evaluated prior to protocol entry by standard of care testing, including EUS, contrast-enhanced helical abdominal CT scan, or MRI. Patients meeting NCCN criteria for potentially resectable (borderline or resectable) tumors will be eligible. Subjects are randomized to receive either 2 cycles of PGH - gemcitabine and nab-paclitaxel (1000 mg/m2 & 125 mg/m2, respectively: days 1, 8, and 15) plus oral HCQ (1200 mg PO daily) - or PGH plus Avelumab (PGHA; days 1 and 15 of each 28-day cycle), by means of response-adaptive randomization based on Grade IIB or greater histologic response.

Surgical exploration and pancreatectomy is performed if technically feasible and all toxicities have resolved. HCQ is taken until the evening before surgery. Avelumab is administered every two weeks until up to one week prior to the date of surgery. The Study Coordinator informs subjects of the date of operation. Following successful surgical removal of tumors, patients are then be free to pursue standard of care adjuvant therapy options, at the discretion of their treating physician.

ELIGIBILITY:
Inclusion Criteria

* Participants with biopsy-proven adenocarcinoma of the pancreas that is determined to be potentially or borderline resectable by NCCN criteria
* Karnofsky performance status of 70-100%
* No active second malignancy with the exception of basal or squamous cell carcinoma of the skin
* Patient has adequate biological parameters as demonstrated by the following blood counts at screening (obtained ≤14 days prior to randomization)

  * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L,
  * Platelet count ≥100,000/mm3 (100 × 109/L),
  * Hemoglobin (Hgb) ≥9 g/dL. Patient may receive transfusion as needed.
* Patient has the following blood chemistry levels at Baseline (obtained ≤14 days prior to randomization):

  * AST (SGOT), ALT (SGPT) ≤ 2.5 × upper limit of normal range (ULN).
  * Total bilirubin ≤ ULN (Except in patients who have Gilbert's Syndrome or patients with recently placed stents for biliary obstruction when bilirubin should be < 1.5 X ULN).
  * Serum Creatinine ≤ 1.5mg/dl OR calculated creatinine clearance ≥ 50 for those patients with creatinine greater than 1.5.
  * CPK < ULN.
  * Patients who have an elevated lipase or amylase and no history of autoimmune pancreatitis, nor physical exam concerning for, or CT correlates of pancreatitis can be enrolled. The elevated levels will serve as the new baseline. Changes above that will be termed toxicities as per CTCAE guidelines with relation to the new baseline.
  * PT WNL+/- 15 % unless on active anticoagulation.
  * PTT WNL+/- 15 % unless on active anticoagulation (suggested to be drawn peripherally to prevent port drawn elevation due to routine heparin flush of ports).
* Age >18 years
* Patient must be able to swallow enteral medications with no requirement for a feeding tube. Patient's must not have intractable nausea or vomiting which prohibits the patient from oral medications
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria

* Subjects deemed surgically unresectable or subjects unwilling to undergo surgical resection
* Prior use of chemotherapy, radiotherapy, and / or investigational agents for pancreatic cancer
* Any evidence of metastasis to distant organs (liver, lung, peritoneum)
* Symptomatic evidence of gastric outlet obstruction
* Inability to adhere to study and/or follow-up procedures
* History of allergic reactions or hypersensitivity to the study drugs (hydroxychloroquine, gemcitabine, nab-Paclitaxel, Avelumab)
* Known or suspected HIV infection
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
  * Patients with controlled Type 1 diabetes mellitus who are on a stable insulin regimen are eligible for the study.
* Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

  * Rash must cover < 10% of body surface area.
  * Disease is well controlled at baseline and requires only low-potency topical corticosteroids.
  * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan
* Patient with a history of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis or pulmonary hypersensitivity pneumonitis

  - History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Active hepatitis B virus (HBV) infection (chronic or acute), defined as having a positive hepatitis B surface antigen (HBsAg) test at screening

  * Patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total hepatitis B core antibody test at screening, are eligible for the study.
  * Active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test followed by a positive HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
* Known clinically significant liver disease, including alcoholic hepatitis, cirrhosis, fatty liver disease, and inherited liver disease
* Active tuberculosis
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 12 months prior to initiation of study treatment, or unstable arrhythmia or unstable angina within 3 months prior to initiation of study treatment
* Grade ≥ 3 hemorrhage or bleeding event within 28 days prior to initiation of study treatment
* Prior allogeneic stem cell or organ transplantation including corneal transplant
* Major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment.

  - Placement of a stent or central venous access catheter (e.g., port or similar) is not considered a major surgical procedure and is therefore permitted.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications as determined by the investigator
* Pregnant or breastfeeding, or intending to become pregnant during the study
* The effects of HCQ, gemcitabine, nab-Paclitaxel and Avelumab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. All females of childbearing potential (please refer to ECOG's definition in section 5.1) must have a blood test or urine study within two weeks prior to randomization to rule out pregnancy. Should a woman become pregnant while participating in this study, she should inform her treating physician immediately. If a man impregnates a woman while participating in this study, he should inform his treating physician immediately as well.
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during treatment with Avelumab or within 5 months after the last dose of Avelumab

  - Attenuated live vaccines include but are not limited to:
* Tuberculosis (BCG)
* Oral polio vaccine
* Measles, Mumps, Rubella, alone or as part of MMR
* Rotavirus
* Yellow Fever
* Typhoid
* Rabies vaccine should be utilized as recommended by an Infectious Disease specialist
* Nasal flu vaccine
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or recombinant human antibodies
* Known allergy or hypersensitivity to any of the study drugs or any of their excipients
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor alpha agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the study, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
  * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection).
* Patients requiring the use of enzyme-inducing anti-epileptic medication that includes but not limited to: phenytoin, carbamazepine, phenobarbital, primidone or oxcarbazepine are excluded
* Patients with previously documented macular degeneration or diabetic retinopathy are excluded
* Baseline EKG with QTc > 470 msec (including subjects on medication). Subjects with ventricular pacemaker for whom QT interval is not measurable will be eligible on a case-by-case basis at MD discretion
* Patients on Coumadin must be willing to switch to an alternative subcutaneous LMWH or oral agent (At PI discretion exceptions can be permitted, as determined on a case by case basis and documented)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Bahary, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PGHA: Gemcitabine, Nab-Paclitaxel, Hydroxychloroquine+Avelumab: Gemcitabine, Nab-Paclitaxel, and hydroxychloroquine and Avelumab
  Days 1, 8, 15 of Cycles 1 and 2: gemcitabine (1000mg/m^2) and nab-paclitaxel (125mg/m^2) Beginning on Day 8 of Cycle 1: hydroxychloroquine (600mg/BID) daily until day of surgery Day 1 of Cycle 3: avelumab (10mg/kg)
- PGH: Gemcitabine, Nab-Paclitaxel, and Hydroxychloroquine: Gemcitabine, Nab-Paclitaxel, and hydroxychloroquine
  Days 1, 8, 15 of Cycles 1 and 2: gemcitabine (1000mg/m^2) and nab-paclitaxel (125mg/m^2) Beginning on Day 8 of Cycle 1: hydroxychloroquine (600mg/BID) daily until day of surgery
Period: Overall Study
Arm/Group | PGHA: Gemcitabine, Nab-Paclitaxel, Hydroxychloroquine+Avelumab | PGH: Gemcitabine, Nab-Paclitaxel, and Hydroxychloroquine
Started | 16 | 16
Completed | 15 | 16
Not Completed | 1 | 0
Not completed — Received <1 dose of treatment | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants that received at least one cycle/dose of study treatment.
Groups:
- PGHA: Gemcitabine, Nab-Paclitaxel, Hydroxychloroquine+Avelumab: Gemcitabine, Nab-Paclitaxel, and hydroxychloroquine and Avelumab
  Days 1, 8, 15 of Cycles 1 and 2: gemcitabine (1000mg/m^2) and nab-paclitaxel (125mg/m^2)
  Beginning on Day 8 of Cycle 1: hydroxychloroquine (600mg/BID) daily until day of surgery
- Total: Total of all reporting groups
Arm/Group | PGHA: Gemcitabine, Nab-Paclitaxel, Hydroxychloroquine+Avelumab | PGH: Gemcitabine, Nab-Paclitaxel, and Hydroxychloroquine | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The Safety Cohort includes the 31 participants who received at least one dose. The Efficacy Cohort includes 18 of the 31 participants who received at least one dose, who underwent surgery.
  years
    Safety cohort | 64.4 (6.5) | 69.9 (9.8) | 67.0 (8.7)
    Efficacy cohort: number analyzed (Participants) | 8 | 10 | 18
    Efficacy cohort | 62.2 (6.4) | 65.6 (9.7) | 64.1 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Safety cohort includes the 31 participants who received at least one dose.
  The Efficacy cohort includes 18 of the 31 participants who received at least one dose, who underwent surgery.
  Participants
    Safety cohort: Female | 6 | 7 | 13
    Safety cohort: Male | 9 | 9 | 18
    Efficacy cohort: number analyzed (Participants) | 8 | 10 | 18
    Efficacy cohort: Female | 3 | 5 | 8
    Efficacy cohort: Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Safety cohort includes the 31 participants who received at least one dose. The Efficacy cohort includes 18 of the 31 participants who received at least one dose, who underwent surgery.
  Participants
    Safety cohort: American Indian or Alaska Native | 0 | 0 | 0
    Safety cohort: Asian | 0 | 0 | 0
    Safety cohort: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Safety cohort: Black or African American | 0 | 0 | 0
    Safety cohort: White | 15 | 16 | 31
    Safety cohort: More than one race | 0 | 0 | 0
    Safety cohort: Unknown or Not Reported | 0 | 0 | 0
    Efficacy cohort: number analyzed (Participants) | 8 | 10 | 18
    Efficacy cohort: American Indian or Alaska Native | 0 | 0 | 0
    Efficacy cohort: Asian | 0 | 0 | 0
    Efficacy cohort: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Efficacy cohort: Black or African American | 0 | 0 | 0
    Efficacy cohort: White | 8 | 10 | 18
    Efficacy cohort: More than one race | 0 | 0 | 0
    Efficacy cohort: Unknown or Not Reported | 0 | 0 | 0
Karnofsky Performance Status - Safety Cohort [Count of Participants; unit: Participants] — The Karnofsky Performance Scale Index is an assessment tool for functional impairment used to compare effectiveness of therapy and to assess the prognosis in individual patients. It consists of a comprehensive 11-point scale correlating to percentage values ranging from 100% (no evidence of disease, no symptoms) to 0% (death). Lower Karnofsky scores are associated with a poorer prognosis. Population: The Safety Cohort includes the 31 participants who received at least one dose.
  Participants
    number analyzed (Participants) | 14 | 16 | 30
    Safety Cohort - Karnofsky Score of 90 | 6 | 3 | 9
    Safety Cohort - Karnofsky Score of 100 | 8 | 13 | 21
Karnofsky Performance Status - Efficacy Cohort [Count of Participants; unit: Participants] — Measure Description: The Karnofsky Performance Scale Index is an assessment tool for functional impairment used to compare effectiveness of therapy and to assess the prognosis in individual patients. It consists of a comprehensive 11-point scale correlating to percentage values ranging from 100% (no evidence of disease, no symptoms) to 0% (death). Lower Karnofsky scores are associated with a poorer prognosis. Population: The Efficacy Cohort includes 18 of the 31 participants who received at least one dose, who underwent surgery.
  Participants
    number analyzed (Participants) | 7 | 10 | 17
    Efficacy Cohort - Karnofsky Score of 90 | 4 | 1 | 5
    Efficacy Cohort - Karnofsky Score of 100 | 3 | 9 | 12

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Grade IIb or Higher Histolopathologic Responses
Description: Number of grade IIb+lll+lllm+IV+lVm responses / total number of all grade histolopathologic responses. Histoligic appearance will be assess per the Grading System for Pathological Response: Grade I - Characteristic cytologic changes of malignancy present, but little (< 10%) or no tumor cell destruction is evident; Grade II - Characteristic cytologic changes of malignancy; 10% to 90% of tumor cells are destroyed; Grade IIa - Destruction of 10% to 50% of tumor cells; Grade IIb - Destruction of 51% to 90% of tumor cells; Grade III - Few (< 10%) viable-appearing tumor cells are present; Grade IIIm - Sizable pools of mucin present; Grade IV - No viable tumor cells present; Grade IVm - Acellular pools of mucin present.
Time Frame: up to 3 years
Population: Participants that received at least one cycle/dose of study treatment for whom tissue samples were available for histological evaluation using the Grading System for Pathological Response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- PGHA: Gemcitabine, Nab-Paclitaxel, Hydroxychloroquine+Avelumab: Gemcitabine, Nab-Paclitaxel, hydroxychloroquine and Avelumab
  Days 1, 8, 15 of Cycles 1 and 2: gemcitabine (1000mg/m^2) and nab-paclitaxel (125mg/m^2)
  Beginning on Day 8 of Cycle 1: hydroxychloroquine (600mg/BID) daily until day of surgery
  Day 1 of Cycle 3: avelumab (10mg/kg)
Arm/Group | PGHA: Gemcitabine, Nab-Paclitaxel, Hydroxychloroquine+Avelumab | PGH: Gemcitabine, Nab-Paclitaxel, and Hydroxychloroquine
Number analyzed (Participants) | 6 | 8
percentage of participants | 33.3 [4.3 to 77.7] | 50.0 [18.7 to 81.3]
Statistical Analysis 1: Comparison: PGHA: Gemcitabine, Nab-Paclitaxel, Hydroxychloroquine+Avelumab vs PGH: Gemcitabine, Nab-Paclitaxel, and Hydroxychloroquine; Test type: Superiority; p = 0.63, Fisher Exact; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.30 to 6.71]

2. Secondary Outcome: Change in CA19-9 Levels
Description: Levels of CA19-9 (tumor marker) in preoperative and postoperative tissues will be determined. Higher levels of CA19-9 are associated with progressive disease.
Time Frame: Up to 3 years
Population: Participants that received at least one cycle/dose of study treatment for whom tissue samples were available for analysis.
Measure: Mean (95% Confidence Interval); unit: units per milliliter (U/mL)
Arm/Group | PGHA: Gemcitabine, Nab-Paclitaxel, Hydroxychloroquine+Avelumab | PGH: Gemcitabine, Nab-Paclitaxel, and Hydroxychloroquine
Number analyzed (Participants) | 5 | 5
units per milliliter (U/mL) | -0.37 [-0.87 to 0.13] | -0.88 [-1.54 to -0.22]
Statistical Analysis 1: Comparison: PGHA: Gemcitabine, Nab-Paclitaxel, Hydroxychloroquine+Avelumab vs PGH: Gemcitabine, Nab-Paclitaxel, and Hydroxychloroquine; Test type: Superiority; p = 0.13, t-test, 2 sided; Mean Difference (Final Values) = -0.63, 95% CI 2-sided [-1.00 to -0.25], Standard Deviation 0.52

3. Secondary Outcome: Worst Grade of Adverse Event Experienced At Least Possibly Related to Treatment
Description: Percentage of participants that experienced an adverse event at least possibly related to study treatment, by Grade. Adverse events were evaluated per per NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Time Frame: Up to 6 months
Population: Participants that received at least one cycle/dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percetage of participants
Arm/Group | PGHA: Gemcitabine, Nab-Paclitaxel, Hydroxychloroquine+Avelumab | PGH: Gemcitabine, Nab-Paclitaxel, and Hydroxychloroquine
Number analyzed (Participants) | 15 | 16
percetage of participants
  Grade 1 | 6.7 [0.5 to 49.6] | 6.3 [0.5 to 47.8]
  Grade 2 | 40.0 [12.0 to 76.4] | 18.8 [3.5 to 59.6]
  Grade 3 | 40.0 [12.0 to 76.4] | 62.5 [26.0 to 88.8]
  Grade 4 | 6.7 [5.1 to 49.6] | 0.0 [0.0 to 40.9]
  Grade 5 | 6.7 [5.1 to 49.6] | 6.3 [0.5 to 47.8]
  No Adverse Events | 0.0 [0.0 to 52.5] | 6.3 [0.5 to 47.8]

4. Secondary Outcome: Worst Grade of Adverse Event Experienced At Least Probably Related to Treatment
Description: Percentage of participants that experienced an adverse event at least probably related to study treatment, by Grade. Adverse events were evaluated per per NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Time Frame: Up to 6 months
Population: Participants that received at least one cycle/dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PGHA: Gemcitabine, Nab-Paclitaxel, Hydroxychloroquine+Avelumab | PGH: Gemcitabine, Nab-Paclitaxel, and Hydroxychloroquine
Number analyzed (Participants) | 15 | 16
percentage of participants
  Grade 1 | 13.3 [1.8 to 56.0] | 12.5 [1.7 to 54.0]
  Grade 2 | 33.3 [8.9 to 71.9] | 18.8 [3.5 to 59.6]
  Grade 3 | 33.3 [8.9 to 71.9] | 43.3 [14.5 to 78.1]
  Grade 4 | 0.0 [0.0 to 42.4] | 0.0 [0.0 to 40.9]
  Grade 5 | 0.0 [0.0 to 42.4] | 0.0 [0.0 to 40.9]
  No Adverse Events | 20.0 [3.7 to 61.8] | 25.0 [0.6 to 64.7]

5. Secondary Outcome: Autophagy Biomarker Levels by Histopathological Response
Description: Autophagy biomarker levels in blood by histopathological response (per the Grading System for Pathological Response)
Time Frame: Up to 3 years
Population: Collected specimens will not be run/analyzed due to lack of funding.
Arm/Group | PGHA: Gemcitabine, Nab-Paclitaxel, Hydroxychloroquine+Avelumab | PGH: Gemcitabine, Nab-Paclitaxel, and Hydroxychloroquine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Coagulation Index (CI)
Description: Comparison of the preoperative and postoperative Thromboelastogram (TEG) Coagulation Index (CI) profile. TEG is an overall assessment of coagulability, quantitatively measures the ability of whole blood to form a clot. Cancer patients are at greater risk for thromboembolism compared to the normal population due to tumor burden and systemic therapies.
Time Frame: up to 3 years
Population: Collected specimens will not be run/analyzed due to lack of funding.
Arm/Group | PGHA: Gemcitabine, Nab-Paclitaxel, Hydroxychloroquine+Avelumab | PGH: Gemcitabine, Nab-Paclitaxel, and Hydroxychloroquine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months per participant; 18 months for each cohort
Description: All adverse events were graded according to the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.0.
  Serious Adverse Events included only events of Grade 3 or greater.
Arm/Group | PGHA: Gemcitabine, Nab-Paclitaxel, Hydroxychloroquine+Avelumab | PGH: Gemcitabine, Nab-Paclitaxel, and Hydroxychloroquine
All-Cause Mortality (participants affected / at risk) | 1/15 | 1/16
Serious Adverse Events (participants affected / at risk) | 9/15 | 12/16
Other Adverse Events (participants affected / at risk) | 15/15 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PGHA: Gemcitabine, Nab-Paclitaxel, Hydroxychloroquine+Avelumab (N=15) | PGH: Gemcitabine, Nab-Paclitaxel, and Hydroxychloroquine (N=16)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (8) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Cardiac arrest (Cardiac disorders) | 1 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (4) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (8) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (3)
Fever (General disorders) | 1 (4) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (4) | 1 (3)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (3)
Salivary gland infection (Infections and infestations) | 1 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (4)
Alanine aminotransferase increased (Investigations) | 1 (4) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (8) | 1 (3)
Neutrophil count decreased (Investigations) | 3 (12) | 4 (18)
White blood cell decreased (Investigations) | 2 (8) | 1 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (4) | 2 (7)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (4) | 3 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (8) | 2 (6)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (8) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (3)
Hypotension (Vascular disorders) | 1 (4) | 1 (3)
Thromboembolic event (Vascular disorders) | 1 (4) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PGHA: Gemcitabine, Nab-Paclitaxel, Hydroxychloroquine+Avelumab (N=15) | PGH: Gemcitabine, Nab-Paclitaxel, and Hydroxychloroquine (N=16)
Anemia (Blood and lymphatic system disorders) | 10 (60) | 11 (51)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (8) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Cardiac arrest (Cardiac disorders) | 1 (4) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (3)
Sinus bradycardia (Cardiac disorders) | 2 (16) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 1 (3)
Blurred vision (Eye disorders) | 0 (0) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (4) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (8) | 1 (3)
Diarrhea (Gastrointestinal disorders) | 6 (24) | 4 (12)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (4) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 (12) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (40) | 4 (15)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (3)
Vomiting (Gastrointestinal disorders) | 5 (24) | 1 (6)
Chills (General disorders) | 3 (12) | 0 (0)
Edema limbs (General disorders) | 1 (4) | 2 (6)
Fatigue (General disorders) | 5 (20) | 7 (30)
Fever (General disorders) | 7 (36) | 0 (0)
Hypothermia (General disorders) | 1 (4) | 0 (0)
Infusion related reaction (General disorders) | 3 (12) | 0 (0)
Pain (General disorders) | 2 (8) | 3 (9)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (4) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (4) | 1 (3)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (3)
Salivary gland infection (Infections and infestations) | 1 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (4)
Alanine aminotransferase increased (Investigations) | 9 (64) | 4 (12)
Alkaline phosphatase increased (Investigations) | 6 (40) | 3 (12)
Aspartate aminotransferase increased (Investigations) | 10 (60) | 5 (15)
Blood bilirubin increased (Investigations) | 1 (4) | 0 (0)
CPK increased (Investigations) | 4 (20) | 1 (3)
Creatinine increased (Investigations) | 1 (12) | 1 (6)
Lipase increased (Investigations) | 2 (12) | 4 (12)
Lymphocyte count decreased (Investigations) | 5 (32) | 2 (12)
Neutrophil count decreased (Investigations) | 9 (64) | 6 (39)
Platelet count decreased (Investigations) | 8 (40) | 13 (57)
Serum amylase increased (Investigations) | 1 (4) | 0 (0)
Weight loss (Investigations) | 0 (0) | 3 (9)
White blood cell decreased (Investigations) | 9 (60) | 9 (48)
Anorexia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (4) | 3 (10)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (4) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (40) | 6 (33)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (24) | 5 (21)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (20) | 1 (3)
Hyponatremia (Metabolism and nutrition disorders) | 7 (48) | 8 (42)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (4) | 2 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Dizziness (Nervous system disorders) | 2 (8) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (4) | 1 (3)
Lethargy (Nervous system disorders) | 1 (4) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (3)
Anxiety (Psychiatric disorders) | 1 (8) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (4) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (4) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (6)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (20) | 3 (12)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5 (36) | 1 (3)
Hypertension (Vascular disorders) | 1 (4) | 2 (15)
Hypotension (Vascular disorders) | 1 (12) | 2 (6)
Thromboembolic event (Vascular disorders) | 1 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT03344172/Prot_SAP_000.pdf